CLINICAL TRIAL: NCT01138436
Title: A Phase II, Randomized, Controlled, Two-Center Pilot Study of the Safety and Efficacy of Topically Applied MEBO® Wound Ointment Compared to Standard of Care in Subjects With Venous Leg Ulcers
Brief Title: A Clinical Study of the Safety and Efficacy of MEBO Wound Ointment in Subjects With Venous Leg Ulcers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Skingenix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEBO-VSU-PII-001 v2.0
Record Dates: First submitted 2010-06-04; First posted 2010-06-07 (Estimated); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Ulcers
Keywords: Venous Leg Ulcers, VLU
MeSH Terms: conditions — Ulcer | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MEBO Wound Ointment (MEBO) (Experimental): Topical application once a day
  Interventions: Drug: MEBO Wound Ointment (MEBO)
- Standard of Care (Active Comparator): Application of Profore multilayer compression bandage system
  Interventions: Procedure: Standard of Care

INTERVENTIONS:
Drug: MEBO Wound Ointment (MEBO) — Topical application once a day
  Other Names: MEBO
  Arms: MEBO Wound Ointment (MEBO)
Procedure: Standard of Care — Application of Profore multilayer compression bandage system
  Arms: Standard of Care

SUMMARY:
This is a Phase II, randomized, controlled, two-center pilot study designed to assess the safety and efficacy of MEBO in the treatment of 14 subjects with VLUs. Subjects meeting entry criteria will be randomly assigned in a 1:1 ratio for up to 8 weeks of treatment with either MEBO or SOC (7 subjects per treatment arm).

DETAILED DESCRIPTION:
To assess the safety and efficacy of MEBO in the treatment of 14 subjects with VLUs. Subjects meeting entry criteria will be randomly assigned in a 1:1 ratio for up to 8 weeks of treatment with either MEBO or SOC (7 subjects per treatment arm).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years of age.
2. Able and willing to provide informed consent.
3. Able and willing to comply with protocol visits and procedures.
4. A full-thickness VLU that has been open continuously for ≥4 weeks and ≤1 year.

Exclusion Criteria:

1. Ulcer of a non-venous hypertensive pathophysiology.
2. Known or suspected allergy to any of the components of MEBO.
3. Malignancy on target ulcer limb.
4. Received another investigational device or drug within 30 days of enrollment.
5. Non-compliance in the screening or run-in period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-11; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Incidence of complete healing of the target ulcer within the 8-week treatment period. | 8 week treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Robert Kirsner, MD, PhD, Study Chair — University of Miami
Locations (2):
- United States (2):
  - Center for Clinical Research, Inc., Castro Valley, California
  - University of Miami Miller School of Medicine, Miami, Florida

IPD SHARING:
Plan to Share IPD: No